CLINICAL TRIAL: NCT04054492
Title: A Randomized, Multi-center, Controlled Clinical Trial for Evaluating the Immunogenicity and Safety of Sequential Immunization Schedules of Sabin IPV and bOPV
Brief Title: To Evaluate the Immunogenicity and Safety of Sequential Immunization Schedules of Sabin IPV and bOPV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Inner Mongolia Autonomous Region Center for Diseases Prevention and Control (Unknown); Shaanxi Provincial Center for Disease Control and Prevention (Other); Hubei Provincial Center for Disease Control and Prevention (Other); Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: sIPV-2018XG-02
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Vaccination; Reaction - Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sIPV+bOPV+bOPV (Experimental): 202 subjects were vaccinated with 1 dose of Sabin-IPV and 2 doses of bOPV at their age of 2/3/4 months old, respectively
  Interventions: Biological: Sabin-IPV+bOPV+bOPV
- sIPV+sIPV+bOPV (Active Comparator): 197 subjects were vaccinated with 2 doses of Sabin-IPV and 1 dose of bOPV at their age of 2/3/4 months old, respectively
  Interventions: Biological: Sabin-IPV+Sabin-IPV+bOPV
- sIPV+sIPV+sIPV (Active Comparator): 205 subjects were vaccinated with 3 doses of Sabin-IPV at their age of 2/3/4 months old, respectively
  Interventions: Biological: Sabin-IPV+Sabin-IPV+Sabin-IPV

INTERVENTIONS:
Biological: Sabin-IPV+bOPV+bOPV — 202 subjects were vaccinated with 1 dose of Sabin-IPV and 2 doses of bOPV at their age of 2/3/4 months old, respectively
  Arms: sIPV+bOPV+bOPV
Biological: Sabin-IPV+Sabin-IPV+bOPV — 197 subjects were vaccinated with 2 doses of Sabin-IPV and 1 dose of bOPV at their age of 2/3/4 months old, respectively
  Arms: sIPV+sIPV+bOPV
Biological: Sabin-IPV+Sabin-IPV+Sabin-IPV — 205 subjects were vaccinated with 3 doses of Sabin-IPV at their age of 2/3/4 months old, respectively
  Arms: sIPV+sIPV+sIPV

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of sequential immunization schedules of Sabin IPV and bOPV.

DETAILED DESCRIPTION:
A phase 4 clinical trial is designed to evaluate the safety and immunogenicity of different sequential immunization schedules of Sabin IPV and bOPV. To be specific, the subjects were divided into 3 groups.

Group 1 received Sabin-IPV+bOPV+bOPV respectively at the age of 2,3,4 months old.

Group 2 received Sabin-IPV+Sabin-IPV+bOPV respectively at the age of 2,3,4 months old.

Group 3 received Sabin-IPV+Sabin-IPV+Sabin-IPV respectively at the age of 2,3,4 months old.

Blood samples were collected before vaccination and 30 days after the third dose. Neutralization antibody against type I, Type II and Type III poliomyelitis virus were detected to evaluate the seroprotection rates and antibody geometric mean concentrations. The safety of the 3 immunization schedule groups were also monitored.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged from 60 days to 89 days old at the date of recruitment;
* with informed consent signed by parent(s) or guardians;
* parent(s) or guardians are able to attend all planned clinical appointments and obey and follow all study instructions;
* subjects did not receive any vaccination within 14 days;
* axillary temperature ≤37.0℃

Exclusion Criteria:

* allergic to any ingredient of vaccine or with allergy history to any vaccine;
* acute febrile disease or infectious disease;
* serious chronic diseases;
* any other factor that makes the investigator determines the subject is unsuitable for this study;

Ages: 60 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 604 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates at both baseline and 30 days after the 3rd vaccination | 4 months
  Determine the seroconversion rates of poliovirus (types I,II,III）at both baseline and 30 days after the 3rd vaccination

SECONDARY OUTCOMES:
Neutralizing antibody titers at both baseline and 30 days after the 3rd vaccination | 4 months
  Measure neutralizing antibody titers against poliovirus type I, II and III at both baseline and 30 days after the 3rd vaccination

OTHER OUTCOMES:
the occurrence of adverse events | 6 months
  analyse the numbers and rates of participants who experience adverse events following immunization

CONTACTS AND LOCATIONS:
Overall Officials: Shaohong Yan, Principal Investigator — Inner Mongolia Autonomous Region Center for Diseases Prevention and Control
Locations (1):
- Inner Mongolia Autonomous Region Center for Diseases Prevention and Control, Hohhot, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan S, Chen H, Zhang Z, Chang S, Xiao Y, Luo L, Zhang Z, Sun L, Chen X, Yang Y, Shi X, Guo Y, Sun Y, Li H, Li N, Han S, Ma M, Yang X. Immunogenicity and safety of different sequential schedules of Sabin strain-based inactivated poliovirus vaccination: A randomized, controlled, open-label, phase IV clinical trial in China. Vaccine. 2020 Sep 11;38(40):6274-6279. doi: 10.1016/j.vaccine.2020.07.042. Epub 2020 Jul 31. PMID 32747216